CLINICAL TRIAL: NCT06950931
Title: Posttranslationally Modified Fetuin-A in the Urine as a Marker for Rejection and Prediction of Graft Function in Renal Transplant Recipients, and Concurrent Correlation of Fetuin-A and Histopalogical Findings of Glomerulopathy in Chronic Kidney Disease Patients.
Brief Title: Posttranslationally Modified Fetuin-A in Urine as a Marker for Renal Dysfunction (Patients With Chronic Kidney Disease - With or Without Kidney Transplantation).
Acronym: (uPTM-FetA)
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Martin (Other)
Responsible Party: Principal Investigator, Matej Vnucak, deputy head of Transplant-nephrology Department, University Hospital, Martin
Other Study IDs: TNO_UNM2; grant UK /3030 /2024 (Other Grant/Funding Number: Comenius University in Bratislava)
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-06

CONDITIONS: Transplant Recipient (Kidney); Primary Kidney Transplantation
Keywords: kidney transplant recipient; Urinary post-translationally modified fetuin A; graft failure; acute kidney injury; biopsy of native kidney
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- pacient with or without kindey transplantation: Adult kidney recipients at least 12 months after kidney transplantation (living donor or donor after brain death) with full immunosuppression (calcineurin inhibitors, mycophenolic acid analogues and corticosteroids). Patients undergo indication or protocolar biopsy and provide a sample of the first-morning urine.
  Patients with chronic kidney disease or acute kidney injury who has undergone a kidney biopsy.
  Interventions: Diagnostic Test: uPTM-FeA

INTERVENTIONS:
Diagnostic Test: uPTM-FeA — In this monocentric prospective cohort study, we will measure uPTM-FeA by enzyme-linked immunosorbent assay (ELISA) kit DNLite IVD 103 in cooperation with PromedeusLab. Human uPTM3-DKD ELISA is a colourimetric immunoassay for quantitatively determining human unique Fetuin-A with specific post-translational modification (PTM) in urine.

SUMMARY:
Kidney transplantation is the preferred treatment method for patients with chronic kidney disease. Standard parameters (estimated glomerular filtration, albuminuria) of renal function detection are limited by many factors, therefore they are considered insufficient. Urinary post-translationally modified fetuin A (uPTM-FeA) appears to be a promising biomarker for the early detection of impaired renal function. Increased values were detected in patients with diabetic kidney disease, acute kidney injury and interstitial fibrosis/tubular atrophy.

Patients after kidney transplantation will be included in our analysis, in which the value of uPTM-FeA at the time of kidney graft biopsy performing (indication/ protocolar) and 6th months after biopsy. The study will also include the patients with chronic kidney disease after renal biopsy, when the value of uPTM-FeA be examined and then 6 months after renal biopsy. The analysis will be correlated with the basic characteristics of the donor and recipient, with the results of protocol or indication biopsy, rejection, level and dose of immunosuppression and parameters detecting renal function. The analysis will be correlated with the histopatology result of kidney biopsy.

The study also include patients with chronic kidney disease or acute kidney injury, who undergo renal biopsy. The value of uPTM-FeA be examined at the time of kidney biopsy and then 6 months after and correlated with the basic laboratory parametres and the results biopsy.

The aim of our study is to confirm the reliability of uPTM-FeA as a marker of kidney graft failure with the perspective of including uPTM-FeA examination in routine examination methods. Early detection of kidney graft failure can help save not only the graft, but also prolong the patient's life. And the second aim is correlated the value of uPTM-FeA with the severity of acute kindey injury and diagnosis of chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria for patients with kidney transplatation:

* patient age > 18 years,
* primary kidney transplantation;
* at least 12 months after kidney transplantation;
* immunosuppression: calcineurin inhibitors, mycophenolic acid analogues and corticosteroids;
* living donor or donation after brain death (DBD) donor;
* patient cooperation;
* regular check-ups in Transplant-Nephrology surgery at University Hospital Martin;
* provision of a sample of the first-morning urine;
* signed informed consent.

Exclusion Criteria with kidney transplatation:

* • patient age < 18 years;

  * secondary/tertiary kidney transplantation;
  * kidney transplantation in the last 12 months;
  * absence of ≥1 of the basic immunosuppressants (calcineurin inhibitors, mycophenolic acid analogues and corticosteroids);
  * contaminated sample of the first-morning urine (for example, menstruation);
  * non-provision of a sample of the first-morning urine;
  * disagreement of the patient with the Examination and inclusion in the study.

Inclusion Criteria for patients without kidney transplatation:

* patient age > 18 years,
* chronic kidney injury or acute kidney injury
* performed renal biopsy
* patient cooperation;
* regular check-ups in Transplant-Nephrology surgery at University Hospital Martin;
* provision of a sample of the first-morning urine;
* signed informed consent.

Exclusion Criteria with kidney transplatation:

* patient age < 18 years;
* absence of renal biopsy or non-represenantative sample of renal biopsy
* contaminated sample of the first-morning urine (for example, menstruation);
* non-provision of a sample of the first-morning urine;
* disagreement of the patient with the Examination and inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after primary kidney transplantation, whose undergo protocolar or indication graft biopsy.
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
uPTM-FeA as a reliable marker of early detection of kidney graft dysfunction | From enrollment to the end of study at 4 weeks
  The primary end-point of this study is to determine if uPTM-FeA is a reliable marker of early detection of graft function deterioration or graft failure in KTRs in correlation with UACR and eGFR (by CKD-EPI equation) and the context of biopsy-proven acute rejection.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Martin, Martin, Slovakia, Slovakia

IPD SHARING:
Plan to Share IPD: No
It is a monocenter pilot study